CLINICAL TRIAL: NCT02012647
Title: Evaluating Cortical Physiology Following Unilateral and Bilateral Subthalamic Deep Brain Stimulation in Parkinson's Disease
Brief Title: Subthalamic Deep Brain Stimulation (DBS) in Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-2013; 40115065-2 (Other: UF Research and Compliance Number)
Record Dates: First submitted 2013-11-01; First posted 2013-12-16 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Parkinson's Disease
Keywords: parkinson; PD; parkinson disease; parkinson's; parkinson's disease; parkinsons; parkinsons disease; TMS; DBS; transcranial magnetic stimulation; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- People with Parkinsons Disease (Active Comparator): Participants have been diagnosed with Parkinson's Disease, and as recommended by their physicians, have undergone DBS surgery for both sides of the brain. These participants will undergo TMS and motor physiology testing, and results will be compared to participants without Parkinson's Disease.
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS); Procedure: Motor Physiology Testing
- Healthy Controls (Placebo Comparator): These participants do not have Parkinson's Disease, nor have they had DBS surgery, and are a healthy controls. These participants will undergo TMS and motor physiology testing, and results will be compared to participants with Parkinson's Disease.
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS); Procedure: Motor Physiology Testing

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation (TMS) — Participants sit in a chair that looks like one in a dentist's office. A magnetic coil will be placed on the scalp on one side of the head, overlying the brain's motor cortex to stimulate the brain's output to the muscles in the opposite hand. A second magnetic coil will be placed on the scalp of the opposite side. Recordings from both hands will be made using the magnetic coils placed on scalp. Results will be compared for participants with and without Parkinson's Disease.
Procedure: Motor Physiology Testing — Participants will be asked to move their upper and lower limbs while seated in a chair. Wireless EMG sensors placed on arm and leg muscles will record measurements during this procedure. Upper and lower limb testing will be performed separately.

SUMMARY:
The purpose of this study is to examine the brain changes in people with Parkinson's Disease (PD) after they get deep brain stimulation (DBS) surgery, compared with people who do not have Parkinson's Disease. Treatment of Parkinson's disease is often difficult and challenging. Deep brain stimulation is an established surgical treatment that is effective for the treatment of PD, but the details of why it helps are not known. In order to achieve maximum benefits from this treatment, it is important to understand how it changes the brain. Specifically, the investigators will study electrophysiology, which is the study of how the brain conducts electrical messages to the rest of the body. To do this, the investigators will use transcranial magnetic stimulation (TMS), which is a painless and non-invasive procedure. They will also conduct motor physiology experiments of the upper and lower limbs to collect data about skeletal muscle movement. The data from this study will help explain whether the electrical changes in the brain have any relation to the physical benefits patients with Parkinson's Disease sometimes receive from DBS surgery.

DETAILED DESCRIPTION:
Screening evaluation: The Investigators will ask questions to see if the participant qualifies to be in the study. The screening visit will occur up to 4 months before the first study visit, and can be scheduled to occur on the same day as the first study visit. This evaluation will include a review of medical history and clinical findings related to Parkinson's Disease (if applicable). There may be a neurological exam (physical exam). Women of child bearing potential will take a urine pregnancy test. If applicable, the medications currently used to treat Parkinson's Disease symptoms will be reviewed and subjects will be asked to discontinue them for some hours on the days of the study visits. The investigators do not expect concerns or unwanted consequences arising either from discontinuing the Parkinson's Disease medications or turning off the DBS stimulator for the duration of time proposed in the study.

Participants will be studied under 4 conditions, over a span of as few as two days to as long as two months. The four Conditions are : 1) The DBS stimulator will be turned OFF for both sides. 2) The DBS stimulator will be turned ON for the right side. 3) The DBS stimulator will be turned ON for the left side. 4) The DBS stimulator will be turned ON for both sides. The order of these conditions will be picked randomly.

Participants will be asked not to take PD medications for approximately 12 hours prior to the scheduled visit time, and until after the physiological testing.

Healthy controls will be studied on only one occasion, as they do not have DBS.

Tests performed for each study condition:

1. Parkinson's Participants Only: A neurological examination will be performed by administering several clinical scaled. These clinical scales include the Unified Parkinson's Disease Rating Scale (UPDRS), the self-report Parkinson's Disease Quality of life scale (PDQ-39), MMSE instrument for cognitive (or memory) testing, and Beck Depression Inventory (BDI II) for evaluation of mood and depressive symptoms. The PDQ-39, MMSE, and BDI will each only be administered once and therefore will not be repeated at every study visit.
2. The investigators will determine individual motor evoked potential (MEP) thresholds before beginning the study treatment. MEP will be recorded from a muscle located between the right thumb and index finger, and then from the left thumb and index finger. MEP threshold refers to the amount of stimulation to the brain that is required to activate muscle cells enough to appear on an electromyography (EMG), which records electrical potential in muscle through electrodes placed on the skin.
3. The investigators will use TMS to test motor cortex functions. For these tests, participants will sit in a chair that looks like the one at the dentist's office. A magnetic coil will be placed on the scalp on one side of the head, overlying the brain's motor cortex to stimulate the brain's output to the muscles in the opposite hand. A second magnetic coil will be placed on the scalp of opposite side. Recordings from both hands will be made using the magnetic coils placed on scalp.
4. The investigators will collect data about the muscles of both the upper and lower limbs with a wireless EMG procedure. To do this, small wireless sensors will be placed on the skin over both arm and leg muscles. Participants will be asked to sit in a chair and perform movements with the upper and lower limbs while the EMG records measurements about movement activity. This procedure will be conducted separately for the upper and lower limbs.
5. Participants who have provided consent will be videotaped during the visits.
6. Side effects and adverse events pertaining to this study will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Diagnosis of Parkinson's Disease with bilateral subthalamic nucleus (STN) DBS

Exclusion Criteria:

* Cardiac pacemakers
* Need for diathermy
* Repeat MRI scanning
* Anticoagulant therapy
* Previous neuro surgical procedure or ablative therapy
* Frank dementia according to cognitive screening
* History of seizures
* Pregnancy
* Presence of a terminal illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Motor Cortex Excitability | As few as 1 days and up to 4 months
  We will measure Motor Cortex Excitability by examining circuitries of inhibition found in the motor cortex which have a reduced function in Parkinson's Disease.

SECONDARY OUTCOMES:
Relation between Unified Parkinson's Disease Rating Scale outcomes and physiological measures | As few as 2 days and up to 4 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is used by neurologists to rate the motor impairment of people with Parkinson's Disease. The rater obtains the score by observation and questioning the participant. Higher scores represent greater impairment and scores range from 0-108.
  The data collected from the UPDRS will be compared to physiological data collected with EMG during limb movement tasks. These tasks are used to gather data about skeletal muscle movements. The EMG data will be evaluated individually with an EMG paradigm considering velocity of movement and both antagonist and agonist burst patterns.
Transcallosal Pathway Excitability | As few as 2 days and up to 4 months
  The investigators will examine the effects of unilateral and bilateral stimulation on the excitability of transcallosal pathway, using specific parameters of Transcranial Magnetic Stimulation (TMS).
Physiological Measures | One day
  Physiological data will be collected from healthy controls with EMG during limb movement tasks. These tasks are used to gather data about skeletal muscle movements. The EMG data will be evaluated individually with an EMG paradigm considering velocity of movement and both antagonist and agonist burst patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, MD, Principal Investigator — University of Florida Center for Movement Disorders and Neurorestoration
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: UF Center for Movement Disorders & Neurorestoration — http://movementdisorders.ufhealth.org/